CLINICAL TRIAL: NCT00644540
Title: A Phase II, Observer-Blind, Parallel Groups, Single Center, Extension Study to Evaluate the Immunogenicity and Safety Following a Single Intramuscular Dose of Influenza Vaccines in Healthy Children Who Received Either One or the Other Vaccine in the Previous V70P2 Study.
Brief Title: Immunogenicity and Safety Following a Single Dose of Influenza Vaccines in Healthy Children Who Received Either One or the Other Vaccine (an Adjuvanted Sub-unit Influenza Vaccine and a Non-adjuvanted Split Virion Influenza Vaccine) in the Previous V70P2 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P2E1
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2014-01

CONDITIONS: FLU
Keywords: Influenza; vaccines; children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Influenza Trivalent Inactivated Vaccines
- 2 (Active Comparator)
  Interventions: Biological: Influenza Trivalent Inactivated Vaccines

INTERVENTIONS:
Biological: Influenza Trivalent Inactivated Vaccines — This phase II, observer-blind, parallel groups, single center, extension study will be performed over a period of approximately 6 months in a study population of healthy children up to 48 months of age.
  Up to two hundred and forty-four children (244) having previously participated in Novartis Vaccines Study V70P2 will be vaccinated with the same influenza vaccines received in the previous trial.
  Each subject will receive a single vaccine dose of 0.25mL, or of 0.5mL, if aged respectively up to 35 months or 36 up to 48 months, administered intramuscularly (IM) in the deltoid muscle, preferably of the non-dominant arm.
  Arms: 1
Biological: Influenza Trivalent Inactivated Vaccines — This phase II, observer-blind, parallel groups, single center, extension study will be performed over a period of approximately 6 months in a study population of healthy children up to 48 months of age.
  Up to two hundred and forty-four children (244) having previously participated in Novartis Vaccines Study V70P2 will be vaccinated with the same influenza vaccines received in the previous trial.
  Each subject will receive a single vaccine dose of 0.25mL, or of 0.5mL, if aged respectively up to 35 months or 36 up to 48 months, administered intramuscularly (IM) in the deltoid muscle, preferably of the non-dominant arm.
  Arms: 2

SUMMARY:
The purpose of this research is to evaluate the immunogenicity of a single dose of Influenza Vaccines (0.5mL or 0.25mL) in healthy children aged up to 35 months or 36 up to 48 months. To evaluate the safety and tolerability of a single 0.25mL IM of injection influenza vaccines in healthy children aged up to 35 months; to evaluate the safety and tolerability of a single 0.50mL IM injection of influenza vaccines in healthy children aged up to 48 months.

ELIGIBILITY:
Inclusion Criteria:

* children up to 48 months of age, who received both doses of one of the two study vaccines in the previous V70P2 trial, whose parents/legal guardians have given written informed consent prior to study entry,
* in good health as determined by:medical history, physical examination, clinical judgment of the investigator.

Exclusion Criteria:

* Experience of a severe acute infectious disease in the month prior to study start or experience of a mild acute infection disease in the week prior the study start;
* Any severe acute respiratory disease and infection requiring systemic antibiotic or antiviral therapy ongoing or resolved within 15 days prior to study start (chronic antibiotic therapy for urinary tract prophylaxis is acceptable);
* Fever (defined as axillary temperature ≥ 38.0°C/rectal temperature ≥ 38.5°C) within the 7 days before enrolment;
* Any serious disease including, for example:cancer,autoimmune disease (including rheumatoid arthritis),diabetes mellitus,chronic pulmonary disease,acute or progressive hepatic disease,acute or progressive renal disease;
* Known or suspected impairment/alteration of immune function, for example, resulting from:receipt of immunosuppressive therapy (corticosteroid - except topical or inhaled steroids - or cancer chemotherapy),receipt of immunostimulants,receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study,high risk for developing an immunocompromising disease;
* Bleeding diathesis;
* History of hypersensitivity to any component of the study medication or chemically related substances;
* History of any anaphylaxis, serious vaccine reactions, or allergy to eggs, egg products or any other vaccine component;
* Laboratory confirmed influenza disease in the past 6 months;
* Surgery planned during the study period;
* Receipt of another investigational vaccine or any investigational agent within 30 days prior to study start. All routine vaccines should be given according to local recommendations: routine vaccines or any other vaccines not foreseen in the protocol can be given after the active trial phase (i.e. 4 weeks after last vaccination in the respective season) has been concluded;
* Participation to another trial of an investigational agent within 90 days of enrolment;
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 16 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of a single 0.25mL or 0.5mL IM injection of two different influenza vaccines, in terms of post-immunization geometric mean titers (GMTs), as measured by HI test, in healthy children aged up to 48 months. | 181 days

SECONDARY OUTCOMES:
Immunogenicity of a single 0.25 or 0.5mL IM injection of two different influenza vaccines in terms of seroprotection, and seroconversion or significant increase, as measured by HI test in healthy children aged up to 48 months. | 181 days
To evaluate the safety and tolerability of a single 0.25 or 0.5 mL IM injection of two different influenza vaccines in healthy children aged up to 48 months | 181 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis
Locations (1):
- University of Tampere Medical School, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Result] Vesikari T, Groth N, Karvonen A, Borkowski A, Pellegrini M. MF59-adjuvanted influenza vaccine (FLUAD) in children: safety and immunogenicity following a second year seasonal vaccination. Vaccine. 2009 Oct 23;27(45):6291-5. doi: 10.1016/j.vaccine.2009.02.004. PMID 19840662